CLINICAL TRIAL: NCT07214623
Title: i-ED COIL Use for Reduction of Chronic Subdural Hematoma Post Market Study
Brief Title: Prospective Multi-center Single Arm Study for Subjects With Chronic Subdural Hematoma Treated With i-ED COILs, Either Alone or in Combination With Burr-holes or Mini-craniotomy
Acronym: iCURE cSDH
Status: Not yet recruiting | Type: Observational
Sponsor: Kaneka Medical America LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CLIN-002
Record Dates: First submitted 2025-10-02; First posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Chronic Subdural Hematoma; cSDH; Chronic Subdural Hematomas
MeSH Terms: conditions — Hematoma, Subdural, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Neuro endovascular embolic coil — i-ED COIL, Kaneka Corporation
  Other Names: Embolization coil

SUMMARY:
All participants will be asked to have a minimally invasive procedure for the treatment of chronic subdural hematoma, a blood clot on the brain. Depending on the specific condition patients may also have a surgical procedure, a mini-craniotomy or burr holes where the skull is pierced and the blood clot is drained.

ELIGIBILITY:
Inclusion Criteria:

* Pre morbid mRS 0-3
* Chronic subdural symptomatic, requiring intervention

Exclusion Criteria:

* Acute subdural hematoma
* Intercranial mass other than subdural hematoma
* Females pregnant or breast feeding
* Compromised survival or inability to complete trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic subdural hematomas with symptoms
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness | 6 months
  Incidence of hematoma recurrence or progression requiring repeat embolization within 180 days
Safety | 90 days
  Modified rankin scale at 90 days post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Fawaz Al-Mufti, MD, Principal Investigator — Westchester Medical Center; Jan-Karl Burkhardt, MD, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - Westchester Medical Center, Valhalla, New York
  - University of Pennslyvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided